CLINICAL TRIAL: NCT05076422
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Subcutaneous Doses of BI 3006337 in Healthy Male Subjects (Single-blind, Partially Randomised Within Dose Groups, Placebo-controlled, Parallel (Sequential) Group Design)
Brief Title: A Study to Test How Well Men Tolerate Different Doses of BI 3006337
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1466-0001; 2020-002600-38 (EudraCT Number)
Record Dates: First submitted 2021-10-05; First posted 2021-10-13 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- BI 3006337 0.2 mg (Experimental): Solution for subcutaneous (s.c) injection containing 0.2 milligrams (mg) of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 0.5 mg (Experimental): Solution for subcutaneous (s.c) injection containing 0.5 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 1 mg (Experimental): Solution for subcutaneous (s.c) injection containing 1 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 2 mg (Experimental): Solution for subcutaneous (s.c) injection containing 2 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 4 mg (Experimental): Solution for subcutaneous (s.c) injection containing 4 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 8 mg (Experimental): Solution for subcutaneous (s.c) injection containing 8 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 15 mg (Experimental): Solution for subcutaneous (s.c) injection containing 15 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 30 mg (Experimental): Solution for subcutaneous (s.c) injection containing 30 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 50 mg (Experimental): Solution for subcutaneous (s.c) injection containing 50 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 100 mg (Experimental): Solution for subcutaneous (s.c) injection containing 100 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- BI 3006337 150 mg (Experimental): Solution for subcutaneous (s.c) injection containing 150 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: BI 3006337
- Placebo (Placebo Comparator): This arm comprises all placebo-treated participants in the trial who were equally distributed across dose groups. Solution for subcutaneous (s.c) injection of placebo was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 3006337 — BI 3006337
  Arms: BI 3006337 0.2 mg; BI 3006337 0.5 mg; BI 3006337 1 mg; BI 3006337 100 mg; BI 3006337 15 mg; BI 3006337 150 mg; BI 3006337 2 mg; BI 3006337 30 mg; BI 3006337 4 mg; BI 3006337 50 mg; BI 3006337 8 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics of BI 3006337 in healthy male subjects following subcutaneous administration of single-rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Temperature, blood pressure (BP), pulse rate (PR)), 12-lead ECG, and clinical laboratory tests
* Age of ≥18 to ≤55 years at screening (SCR)
* BMI of ≥20.0 to <32.0 kg/m2 at SCR
* A minimum absolute body weight (BW) of 70 kilograms (kg) at SCR
* Male subjects who meet any of the following criteria from the administration of trial medication until 30 days after administration of trial medication:

  * Use of adequate contraception, e.g. any of the following methods (of female partners) plus condom or sexually abstinence (if lifestyle-related): implants, injectables, vaginal contraceptives, intrauterine device, oral contraception (failure rate <1%). In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
  * Surgically sterilised/vasectomised (including hysterectomy with or without bilateral salpingectomy or bilateral oophorectomy of female partner. In case of salpingectomy or oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment).
  * Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea.
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Female gender
* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* 3 times repeated measurement of systolic BP outside the range of 90 to 150 mmHg, diastolic BP outside the range of 50 to 90 mmHg, or PR outside the range of 40 to 100 bpm. In case of documented white coat hypertension the decision for eligibility is left to the investigator.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters Alanine Transaminase (ALT) (1.25xupper limit of normal (ULN)), Aspartate Transaminase (AST) (1.25xULN) and Total Bilirubin (T-BIL) (1.5xULN) or renal parameters (creatinine 1.25xULN) exceeding the Upper Limit of Normal (ULN) as specified: after 2 times repeated measurements
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections, including positive tests for Hepatitis (Hep) B antigen/ Hep C antibodies, Human immunodeficiency virus (HIV)-1/2 antibodies and Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- SGS Life Science Services - Clinical Research, Edegem, Belgium
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-blind, partially randomized within dose groups, placebo-controlled, single rising dose, parallel (sequential) group study in healthy male participants.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | BI 3006337 0.2 mg | BI 3006337 0.5 mg | BI 3006337 1 mg | BI 3006337 2 mg | BI 3006337 4 mg | BI 3006337 8 mg | BI 3006337 15 mg | BI 3006337 30 mg | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Started | 19 | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9
Completed | 19 | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were entered and treated with any dose of BI 3006337 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 3006337 0.2 mg | BI 3006337 0.5 mg | BI 3006337 1 mg | BI 3006337 2 mg | BI 3006337 4 mg | BI 3006337 8 mg | BI 3006337 15 mg | BI 3006337 30 mg | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg | Total
Number analyzed (Participants) | 19 | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (9.7) | 43.0 (5.4) | 42.7 (6.2) | 44.8 (6.9) | 46.3 (6.5) | 41.6 (8.8) | 44.8 (10.0) | 46.2 (5.3) | 33.0 (14.2) | 41.2 (9.0) | 39.5 (13.9) | 37.2 (12.1) | 41.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 19 | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9 | 78
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 15 | 5 | 5 | 5 | 6 | 5 | 3 | 5 | 4 | 6 | 6 | 9 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events (AEs) After a Single Dose of BI 3006337
Description: Number of subjects with drug-related adverse events (AEs) after a single dose of BI 3006337 is reported. For drug-related adverse events, medical judgment was used to determine whether there was a reasonable possibility of a causal relationship between the AE and the given trial treatment, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.
Time Frame: From 1 day pre-dose till end of trial, up to 40 days
Population: Treated set (TS): The treated set included all subjects who were entered and treated with any dose of the trial drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BI 3006337 0.2 mg | BI 3006337 0.5 mg | BI 3006337 1 mg | BI 3006337 2 mg | BI 3006337 4 mg | BI 3006337 8 mg | BI 3006337 15 mg | BI 3006337 30 mg | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 19 | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9
Participants | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 3006337 in Serum Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 3006337 in serum over the time interval from 0 extrapolated to infinity is reported (AUC0-∞).
Time Frame: Within 2 hours (h) before drug intake and at 3, 7, 11, 15, 23, 27, 31, 35, 39, 47, 58, 72, 96, 120, 168, 240, 336, 504, 672 h after drug intake and at Day 36.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects in the TS who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS even if he contributed only one PK parameter value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h‧ng/mL)
Arm/Group | BI 3006337 0.2 mg | BI 3006337 0.5 mg | BI 3006337 1 mg | BI 3006337 2 mg | BI 3006337 4 mg | BI 3006337 8 mg | BI 3006337 15 mg | BI 3006337 30 mg | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9
hour*nanogram per milliliter (h‧ng/mL) | NA (NA) — PK parameter could not be determined as too many samples had below limit of quantification concentrations. | NA (NA) — PK parameter could not be determined as too many samples had below limit of quantification concentrations. | 534 (20.7) | 1200 (52.8) | 2870 (32.5) | 3190 (44.9) | 7920 (26.5) | 15100 (38.4) | 40100 (44.2) | 71300 (37.9) | 80600 (34.6)

3. Secondary Outcome: Maximum Measured Concentration of BI 3006337 in Serum (Cmax)
Description: Maximum measured concentration of BI 3006337 in serum (Cmax) is reported.
Time Frame: as for outcome 2
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects in the TS who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS even if he contributed only one PK parameter value to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ml)
Arm/Group | BI 3006337 0.2 mg | BI 3006337 0.5 mg | BI 3006337 1 mg | BI 3006337 2 mg | BI 3006337 4 mg | BI 3006337 8 mg | BI 3006337 15 mg | BI 3006337 30 mg | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9
nanogram per milliliter (ng/ml) | 1.78 (43.5) | 4.38 (75.1) | 4.70 (34.2) | 14.5 (63.7) | 37.3 (79.3) | 50.8 (18.7) | 127 (42.2) | 220 (37.5) | 642 (49.6) | 788 (63.0) | 1290 (54.6)

4. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of BI 3006337 in Serum (Tmax)
Description: Time from dosing to the maximum measured concentration of BI 3006337 in serum (tmax) is reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (h)
Arm/Group | BI 3006337 0.2 mg | BI 3006337 0.5 mg | BI 3006337 1 mg | BI 3006337 2 mg | BI 3006337 4 mg | BI 3006337 8 mg | BI 3006337 15 mg | BI 3006337 30 mg | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 4 | 5 | 4 | 6 | 6 | 9
hour (h) | 7.0 [7.0 to 27.1] | 15.0 [7.0 to 23.1] | 11.0 [7.0 to 72.0] | 15.0 [7.0 to 35.0] | 11.0 [11.0 to 15.1] | 13.0 [11.0 to 23.2] | 11.0 [7.0 to 11.1] | 13.0 [11.0 to 31.0] | 11.0 [11.0 to 27.0] | 61.5 [11.1 to 96.4] | 11.0 [7.0 to 35.0]

ADVERSE EVENTS:
Time Frame: From 1 day pre-dose till end of trial, up to 40 days
Description: Adverse events were reported for the treated set (TS). The TS included all subjects who were entered and treated with any dose of BI 3006337 or placebo.
Groups:
- BI 0.2mg: Solution for subcutaneous (s.c) injection containing 0.2 milligrams (mg) of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 0.5mg: Solution for subcutaneous (s.c) injection containing 0.5 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 1mg: Solution for subcutaneous (s.c) injection containing 1 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 2mg: Solution for subcutaneous (s.c) injection containing 2 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 4mg: Solution for subcutaneous (s.c) injection containing 4 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 8mg: Solution for subcutaneous (s.c) injection containing 8 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 15mg: Solution for subcutaneous (s.c) injection containing 15 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 30mg: Solution for subcutaneous (s.c) injection containing 30 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 50mg: Solution for subcutaneous (s.c) injection containing 50 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 100mg: Solution for subcutaneous (s.c) injection containing 100 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
- BI 150mg: Solution for subcutaneous (s.c) injection containing 150 mg of BI 3006337 was administered once as a single dose subcutaneously following an overnight fast of at least 10 hours (h) before dosing.
Arm/Group | Placebo | BI 0.2mg | BI 0.5mg | BI 1mg | BI 2mg | BI 4mg | BI 8mg | BI 15mg | BI 30mg | BI 50mg | BI 100mg | BI 150mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/5 | 0/6 | 0/5 | 0/6 | 0/5 | 0/4 | 0/5 | 0/4 | 0/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/5 | 0/6 | 0/5 | 0/6 | 0/5 | 0/4 | 0/5 | 0/4 | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 9/19 | 3/5 | 3/6 | 1/5 | 1/6 | 3/5 | 0/4 | 0/5 | 0/4 | 3/6 | 4/6 | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | BI 0.2mg (N=5) | BI 0.5mg (N=6) | BI 1mg (N=5) | BI 2mg (N=6) | BI 4mg (N=5) | BI 8mg (N=4) | BI 15mg (N=5) | BI 30mg (N=4) | BI 50mg (N=6) | BI 100mg (N=6) | BI 150mg (N=9)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Medical device site irritation (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pustule (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-11-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT05076422/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT05076422/SAP_001.pdf